CLINICAL TRIAL: NCT01335321
Title: Prospective And Randomized Study Evaluating Tthe Effect Of The Association Of Triamcinolone To The Viscosupplementation Of The Knee
Brief Title: Evaluation of the Effect of Adding Corticosteroid to Viscosupplementation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, MD, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2010/11450-9
Record Dates: First submitted 2011-04-12; First posted 2011-04-14 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2011-03

CONDITIONS: Osteoarthritis
Keywords: viscosupplementation; intra-articular injection; hyaluronic acid; osteoarthritis; knee
MeSH Terms: conditions — Osteoarthritis | interventions — hylan; Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hylan GF-20 alone (Active Comparator): This arm will receive a knee infiltration with 6ml of Hylan GF-20 only
  Interventions: Drug: Hylan GF-20 alone
- Triamcinolone (Experimental): This arm will receive a knee infiltration with 6ml of Hylan GF-20 associated with 1ml of triamcinolone
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Hylan GF-20 alone — A intraarticular injection of 6ml of Hylan GF-20 (Synvisc)
  Other Names: Synvisc One
  Arms: Hylan GF-20 alone
Drug: Triamcinolone — A Intraarticular injection of 6ml of Hylan GF-20 (Synvisc) + 1ml of triamcinolone (Triancil)
  Other Names: Synvisc One and Triancil
  Arms: Triamcinolone

SUMMARY:
The purpose of this study is to evaluate if the investigators can achieve better early outcomes adding triamcinolone to the viscosupplementation procedure.

DETAILED DESCRIPTION:
So far there is no convincing evidence that any treatment can be really effective in slowing or preventing the development of OA. The viscosupplementation by intraarticular injection of hyaluronate-derived products has gained popularity as a treatment modality of gonarthrosis. Today there are various papers on the treatment of gonarthrosis by intraarticular injection. Several methods have shown good results. There isn't, however, a consensus on the best method. The investigators know that in the treatment of osteoarthritis, with the viscosupplementation Hylan is superior in the long term, than the infiltration with cortisone. The good short term results achieved by infiltration of cortisone make us think about the combination of these drugs. The investigators will be assessing 104 patients with osteoarthritis of the knee, divided into two groups. Patients in group 1 will be subjected to infiltration procedure 6ml of Hylan. Patients in Group 2 will undergo the procedure of infiltration with 6ml of Hylan and 1ml (20mg) of hexacetonide Triamcinolone. The researcher will apply the informed consent term, the pain visual analog scale (VAS), WOMAC and Lequesne questionnaires. The questionnaires will be answered before infiltration (week zero), one week after the puncture (week 1), four weeks after (week 4) and 12 weeks after (week 12) and 24 weeks after (week 24).

ELIGIBILITY:
Inclusion Criteria:

* age between 45 and 80 years
* Osteoarthritis Diagnosis with radiographic evidence
* absence of previous intraarticular knee fracture
* absence of allergy to Synvisc or Triancil

Exclusion Criteria:

* Development of Pioarthritis
* Failure to attend to the consultations

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2011-03; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Results in WOMAC, Lequesne and VAS scores | 4 weeks
  The outcome will be measured with the WOMAC and LEQUESNE scores, both about quality of life and knee function. The subjects will also use the VAS (VISUAL ANALOGIC SCALE) of pain. The results will be compared between the two groups within 1 week and 4 weeks after the viscosupplementation.

SECONDARY OUTCOMES:
Results in WOMAC, Lequesne and VAS scores after 24 weeks | 24 weeks
  The investigators are also going to compare the results after 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Olavo Pires de Camargo, Prof. Dr., Study Chair — Faculdade de Medicina da Universidade de São Paulo
Locations (1):
- Instituto de Ortopedia e Traumatologia do Hospital das Clínicas da Universidade de São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Ozturk C, Atamaz F, Hepguler S, Argin M, Arkun R. The safety and efficacy of intraarticular hyaluronan with/without corticosteroid in knee osteoarthritis: 1-year, single-blind, randomized study. Rheumatol Int. 2006 Feb;26(4):314-9. doi: 10.1007/s00296-005-0584-z. Epub 2005 Feb 10. PMID 15703953
- [Background] Brander VA, Stadler TS. Functional improvement with hylan G-F 20 in patients with knee osteoarthritis. Phys Sportsmed. 2009 Oct;37(3):38-48. doi: 10.3810/psm.2009.10.1728. PMID 20048527
- [Background] Raman R, Dutta A, Day N, Sharma HK, Shaw CJ, Johnson GV. Efficacy of Hylan G-F 20 and Sodium Hyaluronate in the treatment of osteoarthritis of the knee -- a prospective randomized clinical trial. Knee. 2008 Aug;15(4):318-24. doi: 10.1016/j.knee.2008.02.012. Epub 2008 Apr 21. PMID 18430574
- [Background] Goorman SD, Watanabe TK, Miller EH, Perry C. Functional outcome in knee osteoarthritis after treatment with hylan G-F 20: a prospective study. Arch Phys Med Rehabil. 2000 Apr;81(4):479-83. doi: 10.1053/mr.2000.4432. PMID 10768539
- [Background] Kemper F, Gebhardt U, Meng T, Murray C. Tolerability and short-term effectiveness of hylan G-F 20 in 4253 patients with osteoarthritis of the knee in clinical practice. Curr Med Res Opin. 2005 Aug;21(8):1261-9. doi: 10.1185/030079905X56501. PMID 16083536
- [Background] Bannuru RR, Natov NS, Obadan IE, Price LL, Schmid CH, McAlindon TE. Therapeutic trajectory of hyaluronic acid versus corticosteroids in the treatment of knee osteoarthritis: a systematic review and meta-analysis. Arthritis Rheum. 2009 Dec 15;61(12):1704-11. doi: 10.1002/art.24925. PMID 19950318
- [Background] Bellamy N, Campbell J, Robinson V, Gee T, Bourne R, Wells G. Viscosupplementation for the treatment of osteoarthritis of the knee. Cochrane Database Syst Rev. 2006 Apr 19;2006(2):CD005321. doi: 10.1002/14651858.CD005321.pub2. PMID 16625635
- [Background] Chevalier X, Jerosch J, Goupille P, van Dijk N, Luyten FP, Scott DL, Bailleul F, Pavelka K. Single, intra-articular treatment with 6 ml hylan G-F 20 in patients with symptomatic primary osteoarthritis of the knee: a randomised, multicentre, double-blind, placebo controlled trial. Ann Rheum Dis. 2010 Jan;69(1):113-9. doi: 10.1136/ard.2008.094623. PMID 19304567
- [Background] Conrozier T, Jerosch J, Beks P, Kemper F, Euller-Ziegler L, Bailleul F, Chevalier X. Prospective, multi-centre, randomised evaluation of the safety and efficacy of five dosing regimens of viscosupplementation with hylan G-F 20 in patients with symptomatic tibio-femoral osteoarthritis: a pilot study. Arch Orthop Trauma Surg. 2009 Mar;129(3):417-23. doi: 10.1007/s00402-008-0601-2. Epub 2008 Mar 26. PMID 18365224